CLINICAL TRIAL: NCT00887107
Title: Sorafenib as Adjuvant to Radioiodine Therapy in Non-Medullary Thyroid Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Leiden University Medical Center (Other)
Responsible Party: Johannes Smit, M.D., Ph.D., leiden University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL17727.058.07; P07.109
Record Dates: First submitted 2009-04-22; First posted 2009-04-23 (Estimated); Last update posted 2009-04-23 (Estimated); Status verified 2009-04

CONDITIONS: Thyroid Cancer
MeSH Terms: conditions — Thyroid Neoplasms | interventions — Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- sorafenib (Experimental): 30 patients with non-radioiodine avid differentiated thyroid carcinoma
  Interventions: Drug: Sorafenib (nexavar)

INTERVENTIONS:
Drug: Sorafenib (nexavar) — 6 months therapy with Sorafenib 800 mg/day
  Other Names: nexavar

SUMMARY:
The purpose of this study is to assess whether therapy with Sorafenib reinduces radioiodine uptake in thyroid carcinoma.

DETAILED DESCRIPTION:
Background of the study:

Therapy with radioiodine (RaI) is the only curative therapy in non-medullary thyroid carcinoma. RaI uptake is frequently lost in this disease. Therapy with tyrosine kinase inhibitors may restore the susceptibility to RaI.

Objective of the study:

To investigate whether therapy with the tyrosine kinase inhibitor Sorafenib will increase the accumulation of radioiodine (RaI) and decrease tumor progression in patients with recurrences or metastases of non-medullary thyroid carcinoma with absent or insufficient accumulation of RaI.

Study design:

Prospective, open study with patients with recurrences or metastases of differentiated thyroid carcinoma who will undergo 6 months therapy with Sorafenib 800 mg/day. Patients in whom RaI uptake will be restored will be offered high dose (6000 MBq) RaI together with an additional 6 months treatment with Sorafenib. Patients in whom RaI is not be restored but in whom Sorafenib had a favorable effect on tumor growth will be offered continued treatment with Sorafenib.

Study population:

Thirty patients will be included with recurrences or metastases of differentiated thyroid carcinoma that are unresponsive to RaI therapy.

Intervention (if applicable):

After inclusion, patients will undergo 131I scintigraphy as well as a CT scan. Thereafter, therapy with Sorafenib 800 mg/day will be initiated, and continued during 6 months. After 6 months, 131I scintigraphy and CT scans will be repeated. Serum levels of thyroglobulin will be used as tumormarker.

Primary study parameters/outcome of the study:

The endpoint of the study is the proportion of patients with a favorable response to Sorafenib defined as ONE OR MORE of the following criteria:

1. Reinduction of RaI uptake by RaI scintigraphy: The appearance of one or more RaI accumulating lesions at RaI scintigraphy, planar images and/or SPECT (see below)
2. Serum thyroglobulin levels:

   The absence of progression: no statistically significant positive slope at linear regression of the log-transformed serum Tg levels, measured at 0, 4, 8, 12, 16, 20, 24 and 28 weeks after start of Sorafenib:
   * Stable disease: The slope at linear regression of the log-transformed serum Tg levels, measured at 0, 4, 8, 12, 16, 20, 24 and 28 weeks after start of Sorafenib is not significantly different from 0 ln ug/L*time OR
   * Response: The slope at linear regression of the log-transformed serum Tg levels is negative (statistically significantly below 0 ln ug/L*time).
3. CT Imaging:

The absence of progression according to RECIST criteria:

* Stable disease-neither sufficient shrinkage to qualify for partial response nor sufficient increase to qualify for progressive disease, taking as reference the smallest sum longest diameter since the treatment started.
* Partial response-at least a 30% decrease in the sum of the longest diameter of target lesions, taking as reference the baseline sum longest diameter;
* Complete response: the disappearance of all target lesions

ELIGIBILITY:
Inclusion Criteria:

* Patients with non-medullary thyroid carcinoma
* The patients must have undergone total thyroidectomy
* Presence of metastases or inoperable recurrent disease, as proven by elevated serum thyroglobulin levels (Tg) in combination with radiological evidence for tumor
* No or insufficient RaI uptake in tumor as proven by RaI scintigraphy, performed after prior RaI therapy

Exclusion Criteria:

* Pregnancy
* Other active malignancies
* Active kidney, liver or pancreatic disease or dysfunction
* Unstable angina pectoris or recent (<3 months) myocardial infarction.
* Coagulopathy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2007-10

PRIMARY OUTCOMES:
Proportion of patients with a favorable response to Sorafenib defined as ONE OR MORE of the following criteria: 1. Reinduction of RaI uptake by RaI scintigraphy. 2. Serum thyroglobulin levels. 3. RECIST criteria | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Johannes W Smit, MD, PhD, Principal Investigator — Leiden Universty Medical Center
Locations (1):
- Leiden University Medical Center, Leiden, Netherlands

REFERENCES:
- [Derived] Abdulrahman RM, Verloop H, Hoftijzer H, Verburg E, Hovens GC, Corssmit EP, Reiners C, Gelderblom H, Pereira AM, Kapiteijn E, Romijn JA, Visser TJ, Smit JW. Sorafenib-induced hypothyroidism is associated with increased type 3 deiodination. J Clin Endocrinol Metab. 2010 Aug;95(8):3758-62. doi: 10.1210/jc.2009-2507. Epub 2010 May 19. PMID 20484486
- [Derived] Hoftijzer H, Heemstra KA, Morreau H, Stokkel MP, Corssmit EP, Gelderblom H, Weijers K, Pereira AM, Huijberts M, Kapiteijn E, Romijn JA, Smit JW. Beneficial effects of sorafenib on tumor progression, but not on radioiodine uptake, in patients with differentiated thyroid carcinoma. Eur J Endocrinol. 2009 Dec;161(6):923-31. doi: 10.1530/EJE-09-0702. Epub 2009 Sep 22. PMID 19773371